CLINICAL TRIAL: NCT07155200
Title: Small Cell Lung Cancer Irinotecan and CDC2-like Kinase Inhibition Trial (SLICK Trial)
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Biosplice Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 202510135
Record Dates: First submitted 2025-08-26; First posted 2025-09-04 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Small-cell Lung Cancer; Small Cell Lung Carcinoma; Small Cell Lung Cancer
Keywords: Small Cell Lung Cancer; CLK Inhibitors; Cirtuvivint
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Phase I: Irinotecan + Cirtuvivint (Experimental): At the starting dose level, cirtuvivint is administered orally on a 5 days on/2 days off schedule. At all other dose levels (both escalated and de-escalated), cirtuvivint is administered orally on a 2 days/week schedule. Irinotecan is given on Days 1 and 8 of a 21-day cycle at all dose levels
  Interventions: Drug: Cirtuvivint; Drug: Irinotecan
- Phase II: Irinotecan + Cirtuvivint (Experimental): Cirtuvivint is administered orally per the dose and schedule determined in Phase I. Irinotecan is given on Days 1 and 8 of a 21-day cycle.
  Interventions: Drug: Cirtuvivint; Drug: Irinotecan

INTERVENTIONS:
Drug: Cirtuvivint — Cirtuvivint will be supplied by Biosplice.
Drug: Irinotecan — Irinotecan is commercially available.

SUMMARY:
Although small cell lung cancer (SCLC) responds dramatically to initial platinum-based chemotherapy, recurrences are nearly universal. The addition of atezolizumab, an immune checkpoint inhibitor, to front-line chemotherapy has recently demonstrated an improvement in overall survival (OS) in extensive stage SCLC (ES-SCLC). Subsequent lines of therapies are associated with modest efficacy in patients with relapsed disease, and the median overall survival is still 12 to 13 months at best.

Cirtuvivint is a small molecule inhibitor of the CDC2-like kinases (CLKs) and dual-specificity tyrosine-regulated kinases (DYRKs); inhibiting CLKs and DYRKs has been shown in preclinical models to cause tumor growth inhibition and sensitize cancer cells to cytotoxic chemotherapy.

This study is testing the hypothesis that adding cirtuvivint to chemotherapy in patients with relapsed SCLC will be well tolerated and improve the response rate and progression-free survival (PFS).

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed small cell lung cancer that has progressed on at least one line of prior platinum-based chemotherapy, given with or without anti-PD-(L)1 therapy.
* Presence of measurable disease per RECIST 1.1 criteria
* At least 18 years of age.
* ECOG performance status ≤ 2
* Adequate bone marrow and organ function as defined below:

  * Absolute neutrophil count ≥ 1.0 K/cumm
  * Platelets ≥ 100 K/cumm
  * Total bilirubin ≤ 1.5 x IULN
  * AST(SGOT)/ALT(SGPT) ≤ 2.5 x IULN (≤ 5 x IULN for patients with liver metastases)
  * Calculated creatinine clearance > 35 mL/min by Cockcroft-Gault
* The effects of cirtuvivint on the developing human fetus are unknown. For this reason, women of childbearing potential and men must agree to use adequate contraception prior to study entry, for the duration of study participation, and for 31 weeks after completion of study treatment (either drug). Should a woman become pregnant or suspect she is pregnant while participating in this study or should a man suspect he has fathered a child, s/he must inform the treating physician immediately.
* Ability to understand and willingness to sign an IRB approved written informed consent document. Legally authorized representatives may sign and give informed consent on behalf of study participants.

Exclusion Criteria:

* Prior or concurrent malignancy whose treatment or natural history has the potential to interfere with the safety or efficacy assessment of the investigational regimen. Patients with prior or concurrent malignancy that does NOT meet that definition (following discussion with the PI) are eligible for this trial.
* Previous intolerance to irinotecan. Treatment with prior irinotecan is allowed as along as treatment was not discontinued for treatment related adverse events.
* Currently receiving any other investigational agents.
* Patients with untreated symptomatic brain metastases or with clinically evident CNS hemorrhage. Patients with treated brain metastases are allowed if post-treatment brain imaging after CNS-directed therapy shows no evidence of progression. Patients with asymptomatic, punctate brain metastases < 5 mm are allowed.
* A history of allergic reactions attributed to compounds of similar chemical or biologic composition to cirtuvivint, irinotecan, or other agents used in the study.
* Concurrent diarrheal illness (such as inflammatory bowel disease) that requires medical therapy.
* Undergone major surgery within 28 days prior to Cycle 1 Day 1
* Known clinically significant liver disease, including active viral, alcoholic, or other hepatitis, cirrhosis at a level of Child-Pugh B or worse, cirrhosis (any degree) with a history of hepatic encephalopathy or clinically meaningful ascites resulting from cirrhosis (defined as ascites from cirrhosis requiring diuretics or paracentesis), fatty liver, and inherited liver disease.
* Unresolved grade 2 or higher toxicities from previous treatment with the exception of fatigue, lymphopenia, endocrine AEs that are being managed with hormone replacement, alopecia, or dysgeusia.
* Pregnant and/or breastfeeding. Women of childbearing potential must have a negative serum pregnancy test within 7 days prior to C1D1.
* HIV-infected if not on effective anti-retroviral therapy with undetectable viral load for 6 months. Patients with HIV who are receiving effective anti-retroviral therapy and have had an undetectable viral load for at least 6 months are eligible. HIV testing is not required in the absence of known history of infection.
* Evidence of chronic hepatitis B virus (HBV) that is detectable on suppressive therapy. Patients with evidence of chronic HBV infection with undetectable HBV viral load on suppressive therapy are eligible. HBV testing is not required in the absence of known history of infection.
* History of hepatitis C virus (HCV) infection that has not been cured or that has a detectable viral load. Patients with a history of HCV that has been treated and cured are eligible. Patients with HCV infection who are currently on treatment and have an undetectable HCV viral load are eligible. HCV testing is not required in the absence of known history of infection.
* Known retinal abnormalities, including diabetic retinopathy, macular degeneration, other retinal degenerative diseases, or other retinal findings that may place the patient at risk.
* Patients currently using or anticipating the need for food or drugs known to strongly inhibit or induce CYP3A4, such as ketoconazole, itraconazole, erythromycin, or rifampin, within 10 days prior to first dose of study medication.
* Patients with a corrected QT interval (QTc) using Fridericia's formula (QTcF) > CTCAE v5.0 Grade 1 (>480 msec) based on the mean of triplicate evaluation at Screening. In patients with ventricular paced rhythm, a 50 msec subtraction should be applied to the QTc to calculate the QTcF, potential exceptions for patients with pacemakers should be discussed with the PI.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2025-12-18 (Actual); Primary Completion 2028-07-31 (Estimated); Study Completion 2029-01-31 (Estimated)

PRIMARY OUTCOMES:
Recommended Phase II dose (RP2D) (Phase I only) | Through completion of cycle 1 (cycle is 21 days) for all Phase I patients
  - The RP2D is defined as the dose level immediately below the dose level at which 2 patients of a cohort (of 2 to 6 patients) experience dose-limiting toxicity during the first cycle. Dose-limiting toxicities are defined in the protocol.
Objective response rate (ORR) per RECIST criteria (Phase II and RP2D only) | Through completion of treatment (estimated to be 4 months)
  * ORR: Percentage of patients who have a complete response (CR) or partial response (PR).
  * Complete Response (CR): Disappearance of all target lesions. Disappearance of all non-target lesions and normalization of tumor marker level. All lymph nodes must be non-pathological in size (<10 mm short axis).
  * Partial response (PR): At least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters.

SECONDARY OUTCOMES:
Kaplan-Meier Estimate of Progression-Free Survival (PFS) (Phase II and RP2D only) | Through completion of follow-up (estimated to be 10 months)
  * PFS is defined as the duration of time from start of treatment to time of progression or death, whichever occurs first.
  * Progressive Disease (PD): At least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. Appearance of one or more new lesions and/or unequivocal progression of existing non-target lesions. Unequivocal progression should not normally trump target lesion status. It must be representative of overall disease status change, not a single lesion increase.
Kaplan-Meier Estimate of Overall Survival (OS) (Phase II and RP2D only) | Through completion of follow-up (estimated to be 10 months)
  OS is defined as the length of time from start of treatment until date of death.

CONTACTS AND LOCATIONS:
Overall Officials: Ramaswamy Govindan, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu